CLINICAL TRIAL: NCT06730347
Title: A Phase 2 Multicohort Study to Evaluate Lorigerlimab in Participants With Advanced Solid Tumors
Brief Title: A Study of Lorigerlimab in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGD019-03
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Platinum-resistant Ovarian Cancer; Platinum-Resistant Fallopian Tube Carcinoma; Platinum-Resistant Primary Peritoneal Carcinoma; Clear Cell Adenocarcinoma of Ovary; Clear Cell Adenocarcinoma of Vulva; Clear Cell Adenocarcinoma of Vagina; Clear Cell Adenocarcinoma of Cervix; Clear Cell Adenocarcinoma of Uterus; Clear Cell Adenocarcinoma of Fallopian Tube; Clear Cell Adenocarcinoma of Peritoneum; Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PROC Cohort (Experimental): Lorigerlimab IV every 21 days
  Interventions: Biological: Lorigerlimab
- CCGC Cohort (Experimental): Lorigerlimab IV every 21 days
  Interventions: Biological: Lorigerlimab

INTERVENTIONS:
Biological: Lorigerlimab — Bispecific DART protein binding PD-1 and CTLA-4
  Other Names: MGD019

SUMMARY:
Study CP-MGD019-03 is an open-label study of lorigerlimab in participants with platinum-resistant ovarian cancer (PROC) or clear cell gynecologic cancer (CCGC). Approximately 60 participants will be enrolled. The study will assess the efficacy and safety of lorigerlimab in participants with PROC or CCGC.

Participants will receive lorigerlimab by intravenous (IV) infusion on Day 1 of every 21-day treatment cycle. Treatment cycles will continue until progression of cancer, unacceptable side effects, withdrawal of consent by the participant, or the study ends.

Participants will be monitored closely for side effects by physical exam and routine laboratory tests every cycle. Tumor status will be checked approximately every 9 weeks for the first year, then every 12 weeks for the duration of treatment. Participants will have a safety followup performed within 30 days after treatment discontinuation. Participants who discontinue study treatment for reasons other than progression of cancer, will continue CA-125 and tumor assessments every 12 weeks. Participants who discontinue study treatment for progression of cancer will enter the 6-month survival follow up portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high-grade serous epithelial ovarian cancer, including primary peritoneal, or fallopian tube cancer, resistant to platinum based chemotherapy. OR
* Histologically confirmed clear cell carcinoma of the ovary (including primary peritoneal and fallopian tube), endometrium, vagina, vulva, or cervix.
* Persistent or recurrent disease with documented disease progression.
* Participants with PROC must have received at least 1 but not more than 3 prior lines of therapy for PROC.
* Participants with CCGC must have received at least 1 prior line of therapy for CCGC.
* Participants with a known breast cancer (BRCA) mutation (germline or somatic) must have received a a Poly ADP-ribose polymerase (PARP) inhibitor, if locally approved and available, and experienced disease progression or intolerance on the PARP inhibitor.
* Participants must have at least one lesion that meets the definition of measurable disease by RECIST v1.1.
* Participants must have an available archival or formalin-fixed paraffin-embedded tumor tissue, or be willing to undergo a biopsy procedure to obtain a fresh tumor sample.
* Participants have acceptable physical condition and laboratory values.
* Participants of childbearing potential must agree to use highly effective methods of birth control.
* Participants must not be pregnant, planning to be pregnant, or breastfeeding.

Exclusion Criteria:

* Any underlying medical or psychiatric condition impairing participant's ability to receive, tolerate, or comply with the planned treatment or study procedures.
* Primary platinum-refractory disease, defined as disease that did not respond to (CR or PR) or has progressed within 3 months of the last dose of first-line platinum- containing chemotherapy.
* Prior treatment with a checkpoint inhibitor (e.g., anti-PD-1/PD-L1, anti-PD-L2, anti-CTLA-4). Prior use of immune checkpoint inhibitors (e.g., anti-PD-1, anti-PD-L1, anti-CTLA-4) is allowed for clear cell endometrial and clear cell cervical cancer.
* Active brain metastases or leptomeningeal metastases.
* Prior stem cell, tissue, or solid organ transplant.
* Another hematologic or solid tumor ≥ stage 1 malignancy that completed surgery, last dose of radiotherapy, or last dose of systemic anti-cancer therapy ≤ 3 years from first dose of study treatment. Participants with another tumor that has a negligible risk for metastasis or death such as, adequately controlled basal-cell carcinoma or squamous-cell carcinoma of the skin, or carcinoma in situ of the cervix or breast are eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria as determined by the investigator | Throughout the study up to approximately 2 years
  The ORR, is defined as the percentage of patients in the response evaluable population who achieve a best overall response of complete response (CR) or partial response (PR), per RECIST, version 1.1 criteria.
  CR is defined as disappearance of all target and non-target lesions. PR is defined as at least a 30% decrease from baseline in the sum of diameters of target lesions.

SECONDARY OUTCOMES:
Number of participants with adverse event (AEs), serious AEs (SAEs), and AEs leading to study treatment discontinuation. | Throughout the study, up to approximately 2 years
Median duration of response (DoR) per RECIST 1.1 criteria | Throughout the study, up to approximately 2.5 years
  The DoR will be calculated per RECIST v1.1 criteria, as determined by the investigator, from the date of initial tumor response (CR or PR) to the date of first documented progressive disease (PD) or death from any cause, whichever occurs first.
Median progression free survival (PFS) per RECIST 1.1 criteria | Throughout the study, up to 2.5 years
  PFS is defined as the time from the first dose of study treatment to the date of documented PD or death from any cause, whichever occurs first.
Percent change from baseline in tumor size | Throughout the study, up to 2.5 years
  Tumor size is defined as the sum of diameters of the target lesions.
Best percent change from baseline in tumor size | Throughout the study, up to 2.5 years
  Tumor size is defined as the sum of diameters of the target lesions.
Disease control rate (DCR) | Throughout the study, up to 2.5 years
  DCR, per RECIST v1.1 criteria, as determined by the investigator, is defined as the proportion of participants in the response evaluable population who achieve a CR, PR or stable disease for at least 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Pepi Pencheva, Study Director — MacroGenics
Locations (16):
- United States (7):
  - UCLA, Los Angeles, California
  - Ochsner MD Anderson Cancer Center, New Orleans, Louisiana
  - START Midwest, Grand Rapids, Michigan
  - West Penn Allegheny Health, Pittsburgh, Pennsylvania
  - Mays Clinic, Houston, Texas
  - START San Antonio, San Antonio, Texas
  - Wisconsin Institute Medical Research- UW Cancer Connect, Madison, Wisconsin
- Canada (2):
  - Princess Margaret Cancer Center, Toronto, Ontario
  - McGill University, Montreal, Quebec
- South Korea (7):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Hospital Bundang Hospital, Seongnam-si, Gyeonnggi-Do
  - Yonsei University Health System Severance Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No